CLINICAL TRIAL: NCT05362123
Title: Survey the Effectiveness of PLAB Examination in Further Clinical Training in the United Kingdom
Brief Title: Survey on the Effectiveness of the PLAB Examination in Continuing Clinical Education in British Doctors.
Status: Completed | Type: Observational
Sponsor: Jabir Ibn Hayyan Medical University (Other)
Responsible Party: Principal Investigator, Samer Makki Mohamed Al-Hakkak, Head department of Surgery, Jabir Ibn Hayyan Medical University
Other Study IDs: PLAB
Record Dates: First submitted 2022-05-02; First posted 2022-05-05 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: International Medical Graduate Student

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: non interventional — Online google form questioner

SUMMARY:
Online survey for all international medical graduate doctors who decided to get a job in the UK; they must do GMC registration.

ELIGIBILITY:
Inclusion Criteria:

* Post-PLAB exam and GMC registration international medical graduate
* Candidates who practise in NHS as FY1 and FY2

Exclusion Criteria:

* Pass PLAB one exam
* Pass PLAB two exam
* Candidates pass PLAB one and two but still not working in NHS

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: cross-sectional
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-05-03 (Actual); Primary Completion 2022-06-04 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
cross section online google form questioner | 1 month
  cross section online google form questioner

CONTACTS AND LOCATIONS:
Locations (1):
- West Suffolk Hospital, Westbury on Severn, West Suffolk, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided